CLINICAL TRIAL: NCT05207228
Title: Randomized Clinical Trial (RCT) for the Improvement of Cocaine Use Disorder Treatment Through the Implementation of a Cognitive Behavioral Therapy Web-based Treatment (CBT4CBT)
Brief Title: Improvement of Cocaine Use Disorder Treatment Through Cognitive Behavioral Therapy Web-based Treatment (CBT4CBT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-CTB-2020-116
Record Dates: First submitted 2021-04-08; First posted 2022-01-26 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Cocaine Use Disorder
Keywords: Cocaine Use Disorder; Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): After completing the inpatient care (at discharge of inpatient care), patients randomized to TAU will receive day-care / outpatient treatment.
- Treatment as usual + CBT4CBT (Experimental): After completing the inpatient care (at discharge), the patients randomly assigned to the experimental condition will receive the TAU + CBT4CBT a web-based treatment which has been tested on individuals with cocaine use disorder in America by the team of Dr. K.M. Carroll.
  Interventions: Behavioral: CBT4CBT

INTERVENTIONS:
Behavioral: CBT4CBT — Cognitive behavioral treatment through the web CBT4CBT
  Arms: Treatment as usual + CBT4CBT

SUMMARY:
Addictions are among the most serious and expensive public health problems in Europe and Spain and they present high morbimortality. There is an increasing amount of studies emphasizing the role e-health for improving current treatments in mental health but research in addictions is still scarce. Over the last years, there have been several indicators that show an upward trend in the consumption of cocaine and the highly treatment-resistant patients.

Objectives: 1) To evaluate whether adding a web-based cognitive behavioral therapy (CBT4CBT) to standard cocaine use disorder treatment improves treatment outcomes in a Spanish sample of patients with severe addiction 2) To explore differences between men and women in treatment response and psychopathological risk factors of treatment response. Design: Randomized clinical trial. Selection criteria: patients consecutively admitted to the inpatient treatment unit for cocaine detoxification and meet inclusion criteria. Sample: the total sample will be of 70 individuals (randomly assigned to TAU + web-based CBT4CBT (n=35) or to TAU (n=35)). Assessment: Patients will be assessed at the beginning and during inpatient treatment, before and during outpatient treatment (CBT4CBT or TAU), after outpatient treatment (CBT4CBT or TAU) and at follow ups. Treatment retention, changes on craving and related psychological variables as well as presence of benzoylecgonine in urine will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* inpatients for cocaine detoxification in our addiction unit who live in Barcelona or surroundings
* abstinent at the time of the study assessment (from the third day of hospitalization)
* 18 years of age or older.

Exclusion Criteria:

* indication of treatment for reasons other than cocaine detoxification,
* presence of serious psychopathological or neuropsychological alterations that hinder the participation in the study (including severe intoxication)
* opioid abuse or dependence during the last year (this criteria includes maintenance treatment with methadone or another opioid substance)
* a lack of Spanish or Catalan knowledge or difficulties to read or write that hamper the participation in the study,
* Non-acceptance of the study procedures, such as the signing of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Relapse | Through hospitalization completion, an average of 14 days
  Change from baseline at 14 days of inpatient treatment, assessing presence of benzoylecgonine (metabolite of cocaine) in urine after hospitalization and before starting Arm 1 or 2.
Relapse | Through the 8-week period of arm 1 or 2.
  Change from baseline at 8 weeks of outpatient treatment, assessing presence of benzoylecgonine (metabolite of cocaine) in urine during the 8-week period of Arm 1 or 2.
Relapse | At 1 month follow-up after Arm 1 or 2
  Change from baseline at 1 month after outpatient treatment, assessing presence of benzoylecgonine (metabolite of cocaine) in urine at follow-up time point.
Relapse | At 3 months follow-up after Arm 1 or 2
  Change from baseline at 3 months after outpatient treatment, assessing presence of benzoylecgonine (metabolite of cocaine) in urine at follow-up time point.
Relapse | At 6 months follow-up after Arm 1 or 2
  5. Change from baseline at 6 months after outpatient treatment, assessing presence of benzoylecgonine (metabolite of cocaine) in urine at follow-up timepoint.
Treatment retention | Through hospitalization completion, an average of 14 days
  Change from baseline at 14 days of inpatient treatment, after hospitalization and before starting Arm 1 or 2.
Treatment retention | Through the 8-week period of arm 1 or 2
  Change from baseline at 8 weeks of outpatient treatment during the 8-week period of Arm 1 or 2.
Treatment retention | At 1 month follow-up after completing Arm 1 or 2
  Change from baseline at 1 month after outpatient treatment.
Treatment retention | At 3 months follow-up after completing Arm 1 or 2
  Change from baseline at 3 months after outpatient treatment.
Treatment retention | At 6 months follow-up after completing Arm 1 or 2
  Change from baseline treatment retention versus drop out at 6 months after treatment at follow-up time point.

SECONDARY OUTCOMES:
Psychopathology, dependence and craving, as well as anthropometric measures | At baseline, at the beginning of hospitalization
  * MINI international neuropsychiatric interview
  * Symptom CheckList-90 items-Revised. Each dimension has a total score ranging from 0 to 4, where a higher score means higher severity of the symptom.
  * The State-Trait Anxiety Inventory. Every sub-scale has a total score, ranging from 20 to 80, with higher scores correlating with greater anxiety.
  * Beck's Depression Inventory. The total score ranges from 0 to 63, with higher scores indicating a greater severity of the symptoms.
  * Severity of Dependence Scale. The total score ranges from 0 to 15, with a higher score indicating grater dependence.
  * Cocaine Selective Severity Assessment. The scale has a total score ranging from 0 to 126, where a higher score indicates more severity of the withdrawal symptoms.
  * Weiss Cocaine Craving Scale. The total score ranges from 0 to 45, where a higher score indicates more severity of craving symptomatology.
  * Weight is measured in kilograms (Kg)
  * Heigh is measured in meters (m)
Psychopathology, dependence and craving, as well as anthropometric measures | At hospitalization completion, an average of 14 days
  * Symptom CheckList-90 item-Revised. Each dimension has a total score ranging from 0 to 4, where a higher score means higher severity of the symptom.
  * The State-Trait Anxiety Inventory. Every sub-scale has a total score, ranging from 20 to 80, with higher scores correlating with greater anxiety.
  * Beck's Depression Inventory. This instrument has a total score ranging from 0 to 63, with higher scores indicating a greater severity of the symptoms.
  * Severity of Dependence Scale. This questionnaire provides a total score ranging from 0 to 15, with a higher score indicating grater dependence.
  * Cocaine Selective Severity Assessment. The scale has a total score ranging from 0 to 126, where a higher score indicates more severity of the withdrawal symptoms.
  * Weiss Cocaine Craving Scale. The questionnaire has a total score ranging from 0 to 45 where a higher score indicates more severity of craving symptomatology.
  * Weight is measured in kilograms (Kg)
  * Heigh is measured in meters (m)
Psychopathology, dependence and craving, as well as anthropometric measures | Once the 8-week outpatient treatment is completed
  * Symptom CheckList-90 item-Revised. Each dimension has a total score ranging from 0 to 4, where a higher score means higher severity of the symptom.
  * The State-Trait Anxiety Inventory. Every sub-scale has a total score, ranging from 20 to 80, with higher scores correlating with greater anxiety.
  * Beck's Depression Inventory. This instrument has a total score ranging from 0 to 63, with higher scores indicating a greater severity of the symptoms.
  * Severity of Dependence Scale. This questionnaire provides a total score ranging from 0 to 15, with a higher score indicating grater dependence.
  * Cocaine Selective Severity Assessment. The scale has a total score ranging from 0 to 126, where a higher score indicates more severity of the withdrawal symptoms.
  * Weiss Cocaine Craving Scale. The questionnaire has a total score ranging from 0 to 45 where a higher score indicates more severity of craving symptomatology.
  * Weight is measured in kilograms (Kg)
  * Heigh is measured in meters (m)
Psychopathology, dependence and craving, as well as anthropometric measures | At 1 month follow-up after Arm 1 or 2 completion
  * Symptom CheckList-90 item-Revised. Each dimension has a total score ranging from 0 to 4, where a higher score means higher severity of the symptom.
  * Weiss Cocaine Craving Scale. The questionnaire has a total score ranging from 0 to 45 where a higher score indicates more severity of craving symptomatology.
  * Weight is measured in kilograms (Kg)
  * Heigh is measured in meters (m)
Psychopathology, dependence and craving, as well as anthropometric measures | At 3 months follow-up after Arm 1 or 2 completion
  * Symptom CheckList-90 item-Revised. Each dimension has a total score ranging from 0 to 4, where a higher score means higher severity of the symptom.
  * Weiss Cocaine Craving Scale. The questionnaire has a total score ranging from 0 to 45 where a higher score indicates more severity of craving symptomatology.
  * Weight is measured in kilograms (Kg)
  * Heigh is measured in meters (m)
Psychopathology, dependence and craving, as well as anthropometric measures | At 6 months follow-up after Arm 1 or 2 completion
  * Symptom CheckList-90 item-Revised. Each dimension has a total score ranging from 0 to 4, where a higher score means higher severity of the symptom.
  * Weiss Cocaine Craving Scale. The questionnaire has a total score ranging from 0 to 45 where a higher score indicates more severity of craving symptomatology.
  * Weight is measured in kilograms (Kg)
  * Heigh is measured in meters (m)
Addictive behaviors | At baseline, at the beginning of hospitalization
  * South Oaks Gambling Screen. The questionnaire consists of 20 items that lead to a total score, ranging from 0 to 20. As higher is the total score, higher is the probability of pathological gambling.
  * Yale Food Addiction Scale 2. Each item is answered using a 7-point likert scale, ranging from 0 (never) to 7 (always). If the criterion is met, then it is scored as 1. If the score is 0 it means that the criterion has not been met. As more criteria are met, greater is the severity of food addiction.
  * Internet Gambling Disorder (IGM) DSM-5 criteria. As more items are answered as yes, higher is the severity of the internet addiction.
  * Hypersexual Behavior Inventory. Each item is answered using a 5-point likert scale, ranging from 1 (never) to 5 (very often). There are 3 factors and each factor has a total score, so as higher is the score in each factor, higher is the hypersexual behaviour.
Addictive behaviors | Once the 8-week outpatient treatment is completed
  * South Oaks Gambling Screen. The questionnaire consists of 20 items that lead to a total score, ranging from 0 to 20. As higher is the total score, higher is the probability of pathological gambling.
  * Yale Food Addiction Scale 2. Each item is answered using a 7-point likert scale, ranging from 0 (never) to 7 (always). If the criterion is met, then it is scored as 1. If the score is 0 it means that the criterion has not been met. As more criteria are met, greater is the severity of food addiction.
  * Internet Gambling Disorder (IGM) DSM-5 criteria. As more items are answered as yes, higher is the severity of the internet addiction.
  * Hypersexual Behavior Inventory. Each item is answered using a 5-point likert scale, ranging from 1 (never) to 5 (very often). There are 3 factors and each factor has a total score, so as higher is the score in each factor, higher is the hypersexual behaviour.
Personality and emotion regulation | At baseline, at the beginning of hospitalization
  * Sensitivity to Punishment and Sensitivity to Reward Questionnaire. The score of each scale ranges from 0 to 24, with a greater score indicating more sensitivity to punishment or to reward.
  * UPPS-P Impulsive Behaviour Scale. Items are answered using a 4-point likert scale. Each sub-scale has a total score, where high values indicate higher levels of impulsivity.
  * Difficulties in Emotion Regulation Scale. Each item is answered using a 5-point likert scale, and each sub-scale has a total score. As higher is the score in the sub-scale, there are more difficulties in emotional regulation.
  * Emotion Regulation Questionnaire. Items are answered using a 7-point likert scale. Each sub-scale has a total score, where a higher value indicates a greater use of that emotion regulation strategy.
  * Multidimensional Assessment of Interoceptive Awareness. Each item is answered using a 5-point likert scale. There are 8 sub-scales where higher scores indicate higher levels of positive awareness.
Personality and emotion regulation | At hospitalization completion, an average of 14 days
  * UPPS-P Impulsive Behaviour Scale. Items are answered using a 4-point likert scale. Each sub-scale has a total score, where high values indicate higher levels of impulsivity.
  * Difficulties in Emotion Regulation Scale. Each item is answered using a 5-point likert scale, and each sub-scale has a total score. As higher is the score in the sub-scale, there are more difficulties in emotional regulation.
  * Emotion Regulation Questionnaire. Items are answered using a 7-point likert scale. Each sub-scale has a total score, where a higher value indicates a greater use of that emotion regulation strategy.
Personality and emotion regulation | Once the 8-week outpatient treatment is completed
  * UPPS-P Impulsive Behaviour Scale. Items are answered using a 4-point likert scale. Each sub-scale has a total score, where high values indicate higher levels of impulsivity.
  * Difficulties in Emotion Regulation Scale. Each item is answered using a 5-point likert scale, and each sub-scale has a total score. As higher is the score in the sub-scale, there are more difficulties in emotional regulation.
  * Emotion Regulation Questionnaire. Items are answered using a 7-point likert scale. Each sub-scale has a total score, where a higher value indicates a greater use of that emotion regulation strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Núria Mallorquí, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Palazon-Llecha A, Trujols J, Madre M, Duran-Sindreu S, Batlle F, Mallorqui-Bague N. The Predictive Value of Emotion Regulation in Cocaine Use Disorder Severity: Psychotherapeutic Implications During Hospitalization for Detoxification. Clin Psychol Psychother. 2025 Sep-Oct;32(5):e70155. doi: 10.1002/cpp.70155. PMID 40983318
- [Derived] Mallorqui-Bague N, Palazon-Llecha A, Madre M, Batlle F, Duran-Sindreu S, Trujols J. CBT4CBT web-based add-on treatment for cocaine use disorder: Study protocol for a randomized controlled trial. Front Psychiatry. 2023 Mar 2;14:1051528. doi: 10.3389/fpsyt.2023.1051528. eCollection 2023. PMID 36937712